CLINICAL TRIAL: NCT01242644
Title: Comparison of a Pain Pump Versus Injectable Medication for Analgesia in Knee Arthroscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Alabama (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 06-230
Record Dates: First submitted 2010-11-11; First posted 2010-11-17 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Pain Measurement; Ropivacaine; Ketorolac; Morphine; Sulfates

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- pain pump , injectable medication (Experimental): 30mL of ropivacaine (0.5%), 30mg of ketorolac and 8mg of morphine sulfate injected plus a pain pump containing 100mL of ropivacaine (0.5%) administered at 4 mL/hour;
  Interventions: Device: pain pump containing ropivacaine
- saline pain pump , injectable medication (Active Comparator): 30mL of ropivacaine (0.5%), 30mg of ketorolac and 8mg of morphine sulfate injected plus a pain pump containing 100-mL of normal saline administered at 4 mL/hour
  Interventions: Device: saline pain pump with injectable medication
- injectable medication only (Active Comparator): 30mL of ropivacaine (0.5%), 30mg of ketorolac and 8mg of morphine sulfate injected and no pain pump.
  Interventions: Drug: ropivacaine, ketorolac , morphine sulfate

INTERVENTIONS:
Device: pain pump containing ropivacaine — 30mL of ropivacaine (0.5%), 30mg of ketorolac and 8mg of morphine sulfate injected plus a pain pump containing 100mL of ropivacaine (0.5%) administered at 4 mL/hour
  Other Names: ropivacaine; pain; pump
  Arms: pain pump , injectable medication
Device: saline pain pump with injectable medication — 30mL of ropivacaine(0.5%), 30mg of ketorolac and 8mg of morphine sulfate injected plus a pain pump containing 100-mL of normal saline administered at 4 mL/hour
  Other Names: ketorolac; saline
  Arms: saline pain pump , injectable medication
Drug: ropivacaine, ketorolac , morphine sulfate — 30mL of ropivacaine (0.5%), 30mg of ketorolac and 8mg of morphine sulfate injected
  Other Names: morphine; sulfate
  Arms: injectable medication only

SUMMARY:
Hypothesis: Ropivacaine, morphine and ketorolac injected after knee arthroscopy is as effective as this solution plus ropivacaine administered intra-articularly for twenty-four hours.

Three groups were assigned random patients, each group provided a different method of pain medication in order to determine the effectiveness of each treatment.

DETAILED DESCRIPTION:
Arthroscopic knee patients were randomized to 1 of 3 groups. A) 30mL of ropivacaine (0.5%), 30mg of ketorolac and 8mg of morphine sulfate injected plus a pain pump containing 100mL of ropivacaine (0.5%) administered at 4 mL/hour; B) an identical solution plus a pain pump containing 100-mL of normal saline administered at 4 mL/hour; C) an identical solution and no pain pump. Pain level, the amount of pain medication used and time to discharge were recorded. Clinical and radiographic evaluation was performed at nine months after surgery.

ELIGIBILITY:
Inclusion Criteria: All subjects who underwent:

* knee arthroscopy + synovectomy
* knee arthroscopy + partial or complete meniscectomy
* knee arthroscopy + chondroplasty
* knee arthroscopy + microfracture
* knee arthroscopy + autologous osteoarticular transplantation

Exclusion Criteria:

* A surgical procedure that required an incision other then an arthroscopic portal
* A surgical procedure within the same joint within ninety days
* A acute or chronic knee infection
* Any diagnosis of complex regional pain syndrome
* A known allergy to one of the study drugs
* A documented history of narcotic use
* A score of less than two standard deviation on the SF-12 mental component
* Any major systemic or cardiac illness (heart failure, uncontrolled angina, bifascicular blocks, renal insufficiency, or liver disease)
* Under the age of eighteen years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert W Pearsall, MD, Principal Investigator — University of South Alabama

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Started | 16 | 17 | 15
Completed | 16 | 17 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only | Total
Number analyzed (Participants) | 16 | 17 | 15 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (0.9) | 51 (0.9) | 49.9 (0.9) | 51 (0.9)
Sex/Gender, Customized [Number; unit: participants]
  Female | 6 | 10 | 8 | 24
  Male | 10 | 7 | 7 | 24
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 15 | 48

OUTCOME MEASURES:

1. Primary Outcome: Pain Score 8 Hours Post-operativley
Description: Visual Analog Scale. The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain. "no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm).
Time Frame: 8 hours post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Number analyzed (Participants) | 16 | 17 | 15
units on a scale | 2.5 (0.3282) | 1.8 (0.3282) | 1.06 (0.3282)

2. Primary Outcome: Pain Scale
Description: as for outcome 1
Time Frame: 24 hours post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Number analyzed (Participants) | 16 | 17 | 15
units on a scale | 1.75 (0.16) | 3.23 (0.16) | 3.06 (0.16)

3. Primary Outcome: Pain Scale
Description: as for outcome 1
Time Frame: 48 hours post-surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Number analyzed (Participants) | 16 | 17 | 15
units on a scale | 1.81 (0.14) | 3.17 (0.14) | 2.26 (0.14)

4. Primary Outcome: Pain Scale
Description: as for outcome 1
Time Frame: 72 hours post surgery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Number analyzed (Participants) | 16 | 17 | 15
units on a scale | 3.3 (0.46) | 4.05 (0.46) | 3.13 (0.46)

5. Secondary Outcome: Number of Narcotic Pills and Morphine Sulfate Used
Description: Pill count
Time Frame: In recovery room
Measure: Mean (Standard Deviation); unit: Pills
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Number analyzed (Participants) | 16 | 17 | 15
Pills | 2.2 (0.61) | 1.8 (0.61) | 1.3 (0.61)

6. Secondary Outcome: Number of Narcotic Pills and Morphine Sulfate Used
Description: Pill Count
Time Frame: Post surgery day 1
Measure: Mean (Standard Deviation); unit: Number of pills
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Number analyzed (Participants) | 16 | 17 | 15
Number of pills | 3.41 (0.87) | 3.8 (0.87) | 3.8 (0.87)

7. Secondary Outcome: Number of Narcotic Pills and Morphine Sulfate Used
Time Frame: Post surgery day 2
Measure: Mean (Standard Deviation); unit: Number of pills
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Number analyzed (Participants) | 16 | 17 | 15
Number of pills | 1.1 (0.08) | 1.5 (0.08) | 0.8 (0.08)

8. Secondary Outcome: Number of Narcotic Pills and Morphine Sulfate Used
Time Frame: Post surgery day 3
Measure: Mean (Standard Deviation); unit: number of pills
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
Number analyzed (Participants) | 16 | 17 | 15
number of pills | 2.1 (0.16) | 2.7 (0.16) | 1.7 (0.16)

ADVERSE EVENTS:
Time Frame: At 12 months post-operatively
Arm/Group | Pain Pump , Injectable Medication | Saline Pain Pump , Injectable Medication | Injectable Medication Only
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/15
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes